CLINICAL TRIAL: NCT06672302
Title: A Multi-center, Single Arm, Prospective Exploratory in Vitro Diagnostic Devices Clinical Performance Study to Evaluate of in Vitro Diagnostic Devices for Auxiliary Diagnosis That Classifies High-risk and Low Risk Patients With Breast Cancer by Analyzing Surface-enhanced Raman Spectroscopy (SERS) Profiles of Extracellular Vesicles (EVs) Extracted From Human Plasma Using Artificial Intelligence
Brief Title: A Prospective Study to Develop and Clinically Validate an in Vitro Diagnostic Medical Device That Uses Blood to Classify Patients at High Risk for Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: EXoPERT (Industry)
Responsible Party: Sponsor
Other Study IDs: EXP-B-P-2401
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasm
Keywords: Breast; Breast Cancer; Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast malignant nodule group
  Interventions: Diagnostic Test: ExoPred
- Breast benign nodule group
  Interventions: Diagnostic Test: ExoPred

INTERVENTIONS:
Diagnostic Test: ExoPred — Performing in vitro diagnostics with devices developed by EXoPERT

SUMMARY:
EXoPERT has developed a liquid biopsy-based in vitro diagnostic medical device that can diagnose cancer through blood. The in vitro diagnostic medical device for this clinical performance trial is a test device that applies a technology that measures Raman spectroscopic signals of extracellular vesicles in the blood and classifies high-risk and low-risk patients for breast cancer through artificial intelligence analysis.

The test device used in this clinical performance trial is expected to assist in the differential diagnosis of high-risk and low-risk breast cancer patients by developing a software algorithm for an in vitro diagnostic medical device for auxiliary diagnosis that classifies high-risk and low-risk breast cancer patients and confirming the clinical efficacy and safety of the device through this clinical performance trial.

DETAILED DESCRIPTION:
According to the Korean Breast Cancer Society, when comparing the five-year survival rate of breast cancer patients by stage from 2001 to 2012, the survival rate is 98.3% for stage 0, 96.6% for stage 1, and 91.8% for stage 2, but the survival rate for stage 4 patients with systemic metastasis is 34%. Therefore, early detection and accurate diagnosis are very important for breast cancer treatment.

Currently, breast cancer is diagnosed through breast ultrasound and mammography. These imaging modalities are defined by the American College of Radiology's Breast Imaging Reporting and Data System (BI-RADS) to define the specificity and various characteristics of the lesion. BI-RADS is divided into six categories: Category 1 is no abnormality, Category 2 is a definite benign tumor, Category 3 is a high likelihood of benign tumor (≤2% positive predictive value), Category 4 is a low likelihood of malignancy (≤2% positive predictive value), except for Category 0, which is an incomplete determination, Category 4 is a moderate suspicion of malignancy (2< positive predictive value <95%), Category 5 is a very high probability of malignancy (positive predictive value ≥95%), and Category 6 is a pathologically diagnosed malignancy.

In the Breast Imaging Reporting and Data System (BI-RADS), biopsy is not required in category 3 because the likelihood of malignancy is 2% or less, so a 6-month follow-up is recommended, and biopsy is recommended starting from category 4A, where the frequency of malignancy is 3 - 10%. However, the BI-RADS criteria have a significant number of false-positive results, which leads to an increase in unnecessary biopsies. The need for complementary diagnostic tests that can overcome the limitations of conventional imaging tests and compensate for unnecessary biopsies is being emphasized.

ELIGIBILITY:
Inclusion Criteria(Breast malignant nodule group)

1. Korean nationality
2. Voluntary written consent to participate in this clinical performance trial study
3. Confirmed breast cancer through imaging/pathologic diagnostic tests
4. Those who have been diagnosed with breast cancer at a stage prior to treatment and surgery, and who agree to participate in this study and are able to provide blood samples.
5. Those whose lesions have been confirmed by conventional examination (breast ultrasound or mammography) and who fall into BI-RADS categories 4,5,6 and have undergone biopsy or are scheduled to undergo biopsy within 2 weeks.
6. Those who meet the following demographic conditions A. Adult female, 40 years of age or older
7. Those who can provide the following clinical information A. Age and biological sex B. Whether or not they have dense breasts C. Occupational information D. Pathological tumor size, Clinical tumor size, Pathological TNM staging, Clinical TNM staging, tumor location, breast cancer histology findings (breast cancer subtype) E. Family history and past history of cancer F. Breast-related diseases G. Chronic disease history

Inclusion Criteria(Breast benign nodule group)

1. Korean nationality
2. Voluntary written consent to participate in this clinical performance trial study
3. Diagnosed with breast nodules through imaging/pathologic diagnostic tests
4. Those who have been diagnosed with breast nodules and have agreed to participate in this study and are able to provide blood samples at a stage prior to treatment and surgery.
5. Those whose lesions have been confirmed by conventional examination (breast ultrasound or mammography) and fall into BI-RADS categories 4,5,6 and have undergone biopsy or are scheduled for biopsy within 2 weeks
6. Those who meet the following demographic conditions A. Adult female, 40 years of age or older
7. Those who can provide the following clinical information A. Age and biological sex B. Whether or not they have dense breasts C. Occupational information D. Diagnosis, nodule size, and number of nodules E. Family history and past history of cancer F. Breast-related diseases G. Chronic disease history

Exclusion Criteria:

1. Those who have been diagnosed with cancer (malignant tumor) of any type within 5 years of the date of consent and have undergone appropriate chemotherapy/radiation treatment or surgery.
2. Those who are confirmed to have developed breast cancer due to metastasis from malignant tumors other than breast cancer
3. Pregnant women
4. Participation in a drug-related clinical trial within 3 months of the date of the informed consent form

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients categorized as BI-RADS category 4,5,6
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | through study completion, an average of 1 year
Specificity | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided